CLINICAL TRIAL: NCT00542672
Title: Parental Influences on Obesity Among Mexican American Children
Brief Title: Evaluating Parental Influences on Obesity Among Mexican American Children
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1397; R01HL084404-01A2 (NIH)
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Obesity
Keywords: Mexican American; Dietary Intake; Child-Feeding Practices; Weight; Cultural Values
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Latino children in the United States have an increased risk of becoming overweight or obese. Previous studies have suggested that parental behaviors are an important influence on children's weight, but more research is needed on the types of behaviors that may contribute to obesity specifically among Latino children. The purpose of this study is to examine the connection between family eating habits and behaviors and obesity among Mexican-American children.

DETAILED DESCRIPTION:
The number of children in the United States who are overweight or obese has increased steadily over the past several decades. Latino children are at particular risk of becoming overweight or obese. Children who are overweight or obese have an increased risk of high blood pressure, high cholesterol, heart disease, and diabetes. Parental behaviors are thought to be important influences on children's obesity, but previous studies have only examined a narrow range of parental behaviors, and few studies have specifically focused on Latino children. There is an urgent need for further research that examines the ways in which parental eating habits and behaviors affect the rising obesity rates among Latino children. This study will focus on Mexican Americans, which is the largest Latino group in the United States. The purpose of this study is to examine whether parental and extended family members' dietary-related behaviors predict children's dietary intake and weight gain. The effects of socioeconomic status and cultural factors on parental behaviors will also be examined.

This study will enroll Mexican-American children and their parents. All study visits will occur at the participant's home. At a baseline visit, study staff will conduct a 1-hour interview with children and their parents to collect information on their thoughts about food, family eating habits, and how family members talk about food; children will also be asked about their physical development and physical activity level. Both parents and children will have their height, weight, waist, and hip circumference measured. Children will then wear an activity monitor for 3 days in the week following the baseline visit to measure physical activity levels. Two additional study visits will occur over the following 3 weeks. At the second visit, study staff will conduct 20-minute interviews with parents and children about their eating habits. At the third visit, study staff will videotape the child's evening meal, and additional interviews will occur. Follow-up visits will occur at Years 1 and 2. At both follow-up visits, repeat baseline interviews will occur, and children will wear the activity monitor for 3 days.

ELIGIBILITY:
Inclusion Criteria for Children:

* Mexican American
* Age 8 to 10
* Only one child from each family will be eligible to participate; one child will be randomly selected if multiple children are eligible

Inclusion Criteria for Parents:

* Mexican American
* Any marital status
* Speaks Spanish or English
* Family will be eligible to participate even if only mother agrees to participate

Exclusion Criteria for Children:

* Diagnosed with a condition or disease that affects weight (e.g., inflammatory bowel disease, type 1 diabetes, underlying thyroid disease)
* Currently participating in another obesity clinical trial

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mexican American children ages 8-10 whose parent is a member of Kaiser Permanente, an HMO
Sampling Method: Non-Probability Sample
Enrollment: 831 (Actual)
Dates: Start 2008-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Parental and extended family members' dietary-related behaviors and the effect they have on children's dietary intake and weight gain | Measured during study visits at participants' homes

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne M. Tschann, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States